CLINICAL TRIAL: NCT06454942
Title: Impact of Regular Consumption of Eggs and Nutrients Fortified Eggs on Eczema Condition in Singapore Individuals With Eczema
Brief Title: Impact of Regular Consumption of Eggs and Nutrients Fortified Eggs on Eczema Condition in Singapore Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S26
Record Dates: First submitted 2024-04-07; First posted 2024-06-12 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis Eczema; Aging; Diet Modification
Keywords: Atopic Dermatitis; Eczema; Young and Middle-aged adults; Eye health; Antioxidants
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular egg with habitual diet (Experimental): Each subject will be provide one-on-one dietary counselling and written instructions for each subject will be provided by a research dietitian and trained research staff.Subjects will also be provided with 2 regular egg/day for 12 weeks.
  Interventions: Dietary Supplement: Regular egg with habitual diet
- Nutrient-fortified egg with habitual diet (Experimental): Each subject will be provide one-on-one dietary counselling and written instructions for each subject will be provided by a research dietitian and trained research staff.Subjects will also be provided with 2 nutrient-fortified egg/day for 12 weeks.
  Interventions: Dietary Supplement: Nutrient-fortified egg

INTERVENTIONS:
Dietary Supplement: Nutrient-fortified egg — Consumption of nutrient-fortified eggs with habitual diet
  Arms: Nutrient-fortified egg with habitual diet
Dietary Supplement: Regular egg with habitual diet — Consumption of regular egg with habitual diet
  Arms: Regular egg with habitual diet

SUMMARY:
The study aims to assess the effects of daily consumption of nutrients-fortified eggs on eczema condition in Singapore individuals with eczema. The investigators hypothesize that egg consumption will improve eczema condition and nutrients fortified egg consumption will improve further improvements when compared to standard egg consumption in individuals with eczema

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel study and all subjects will complete a 12-week study period. Subjects will be tasked to consume nutrients-fortified eggs and regular eggs daily for 12 weeks. After which, subjects are assessed for changes in carotenoid status, antioxidant and anti-inflammatory biomarkers, skin and eye health measurements, and other biomarkers of health.

ELIGIBILITY:
Inclusion Criteria:

1. English-literate and able to give informed consent in English
2. Male and female participants, aged between 21 and 59 inclusive
3. Healthy individuals with no underlying condition or on regular medication
4. BMI between 18.5-25 kg/m2
5. Mild to moderate severity of eczema, which will also be determined using our questionnaires during the screening visit

Exclusion Criteria:

1. Significant change in body weight (3 kg or more) in the past 3 months
2. Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week
3. Known food allergy to eggs
4. Taking dietary supplements which may impact the study results
5. Having gastrointestinal disorders not suitable for the study
6. Current smokers
7. Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine, 340ml of beer/cider, or 45ml of distilled spirit
8. Taking lipid-lowering and blood pressure-controlling medications for less than 3 years
9. Pregnant or lactating women, or planning to conceive in the next 6 months
10. Unwilling to stop the medication of eczema during the study, either topical creams or oral medications
11. Hierarchical link (professional and familial ties) with the research team members
12. Participating in another clinical study
13. Having blindness in one eye or more, eye diseases, retinal/lens/optical nerve surgery, or other eye conditions that may impact the study results
14. Low-quality macular pigment optical density results were determined during the screening visit.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Skin questionnaires - SCORing Atopic Dermatitis (SCORAD) Index | Week 0, week 3, week 6, week 9, week 12
  SCORing Atopic Dermatitis (SCORAD) Index is a clinical tool used to assess the severity of atopic dermatitis (AD), also known as eczema. This index can estimate participants' body surface area affected by burns (extent - A: percentage of body surface area affected), Intensity (B: clinical signs are assessed and scored on a scale from 0 (absent) to 3 (severe)), Subjective Symptoms (C: itch, sleep disturbance are evaluated based on the participants' report over the past three days, each scored on a scale from 0 (no symptom) to 10(severe symptom)).
  The SCORAD index is calculated using the following formula:
  SCORAD=A/5+7B/2+C
  Interpretation Mild atopic dermatitis: SCORAD < 25 Moderate atopic dermatitis: SCORAD 25-50 Severe atopic dermatitis: SCORAD > 50
Skin questionnaires - Eczema Area and Severity Index (EASI) scoring system | Week 0, week 3, week 6, week 9, week 12
  EASI evaluates the extent and severity of eczema in four body regions: the head and neck, the trunk, the upper limbs, and the lower limbs.
  The EASI score ranges from 0 to 72, with higher scores indicating more severe eczema:
  0: No eczema 1-7: Mild eczema 8-21: Moderate eczema 22-50: Severe eczema 51-72: Very severe eczema
Skin questionnaires - Dermatology life quality index (DLQI) | Week 0, week 3, week 6, week 9, week 12
  DLQI is a dermatology-specific instrument used to measure the impact of skin diseases on patients' quality of life. Which assessed disease impact, monitor treatment effectiveness, guide clinical decision-making.
  Interpretation of Scores:
  0-1: No effect on patient's life 2-5: Small effect on patient's life 6-10: Moderate effect on patient's life 11-20: Very large effect on patient's life 21-30: Extremely large effect on patient's life
Skin measurement - eczema related | Week 0, week 3, week 6, week 9, week 12
  Skin hydration - units arbitrary Corneometer®. Transepidermal water loss - units gram/hour. Sebum level - unit µg/cm2. Skin pH level - skin pH meter. Skin tape stripping: stratum corneum components assessed by immune dot blots
Skin carotenoids status | Week 0, week 3, week 6, week 9, week 12
  Skin carotenoids concentration can be measured by Resonance Raman Spectroscopy, unit is skin carotenoid score, higher score means optimal, lower score means poor condition of skin carotenoids.
Blood carotenoids levels | Week 0, week 6, week 12
  Blood carotenoids levels can be measured by High-Performance Liquid Chromatography, unit is μmol/L.

SECONDARY OUTCOMES:
Eye health - Macular Pigment Optical Density | Week 0, week 3, week 6, week 9, week 12
  A measurement of macular pigment of the eye using a heterochromatic flicker photometry device. The measurements are in arbitrary units.
Eye health - Visual acuity | Week 0, week 3, week 6, week 9, week 12
  Participants will read out letters on a ETDRS LogMAR chart at a fixed distance where letters becomes smaller as it goes down the chart. Tests results will be recorded in number of letters read, where the more letters the better the outcome.
Eye health - Photostress recovery time | Week 0, week 3, week 6, week 9, week 12
  An ophthalmoscope will be used to shine a light into the participants eye for 10 seconds, and participants will be required to read letters off a chart the moment their vision returns to normal. The faster the recovery time, the better the outcome. Units will be in seconds
Visual function questionnaire 25 | Week 0, week 3, week 6, week 9, week 12
  A questionnaire to for participants to self-evaluate their perception of their current eye health based on general vision, ocular pain, near activities, distance activities, vision specific functions, driving, color vision and peripheral vision. The best possible score is 100 and worst possible score is 0.
Concentration of tumour necrosis factor-α | Week 0, week 6, week 12
  The blood obtained from the participants will be processed for storage. Tumor necrosis factor-α results will be presented in ng/L according to the commercially available enzyme-linked immunosorbent assay kits.
Concentration of interleukin-6 | Week 0, week 6, week 12
  The blood obtained from the participants will be processed for storage. Interleukin-6 results will be presented in ng/L according to the commercially available enzyme-linked immunosorbent assay kits.
Concentration of high-sensitivity C-reactive protein | Week 0, week 6, week 12
  The blood obtained from the participants will be processed for storage. High-sensitivity C-reactive protein results will be obtained and presented in mg/L by commercial lab testing.
Concentration of fasting blood glucose | Week 0, week 6, week 12
  Fasting blood glucose will be measured using commercial lab testing using participants' blood, units will be in mmol/L.
Concentration of malondialdehyde | Week 0, week 6, week 12
  The blood obtained from the participants will be processed for storage. Analyses of malondialdehyde using commercially available enzyme-linked immunosorbent assay kits. Units for malondialdehyde will be in ng/L according to assay kit instructions.
Concentration of 8-isoprostaglandin-F2α | Week 0, week 6, week 12
  The blood obtained from the participants will be processed for storage. Analyses of 8-isoprostaglandin-F2α using commercially available enzyme-linked immunosorbent assay kits. Units for 8-isoprostaglandin-F2α will be in µmol/L according to assay kit instructions.
Concentration of insulin | Week 0, week 6, week 12
  Fasting blood insulin will be measured using commercial lab testing using participants' blood, units in μU/L.
Percentage of glycated hemoglobin | Week 0, week 6, week 12
  Glycated hemoglobin will be measured using commercial lab testing from participant's blood, units in percent.
Skin advanced glycation end products levels | Week 0, week 3, week 6, week 9, week 12
  Measurement of skin advanced glycation end products level using a skin autofluorescence device, where participants wlll be instructed to place their forearm over the device and a light will be shone and a reading can be captured by detecting fluorescence. The results will be presented as arbitrary units.
Blood advanced glycation end products levels | Week 0, week 3, week 6, week 9, week 12
  Participants will have their blood drawn by medical professionals at the Occupational Health Clinic. The blood will be processed and stored. Measurements will be done using ultra-performance liquid chromatography coupled with mass spectrometry techniques to determine the levels of advanced glycation end products. Units will be in μg/mL.

OTHER OUTCOMES:
Dietary assessment | Week 0, week 3, week 6, week 9, week 12
  3-day food record will be used to assess participants' dietary intake for two weekdays and one weekend day before each clinical visit.
Measurement of height | Week 0, week 3, week 6, week 9, week 12
  Height will be measured using height-weight scale and units will be in cm.
Measurement of blood pressure | Week 0, week 3, week 6, week 9, week 12
  A blood pressure monitoring device available commercially will be used be to measure their systolic and diastolic blood pressure. Unit is mmHg.
Measurement of weight | Week 0, week 3, week 6, week 9, week 12
  Weight will be measured using height-weight scale and units will be in kg.
Measurement of waist circumference | Week 0, week 3, week 6, week 9, week 12
  Waist circumference will be measured using a measuring tape by a trained personnel, units in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, RD, Principal Investigator — National University of Singapore
Locations (1):
- Department of Food Science and Techonology, Block S13, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The link between participants' information data and the code will be kept confidential by the NUS research team or a trusted third party. Research data and results will only be collated in its coded format. All research data collected will be retained for a minimum of 10 years following the NUS Research Data Management Policy.

REFERENCES:
- [Background] Imai A, Oda Y, Ito N, Seki S, Nakagawa K, Miyazawa T, Ueda F. Effects of Dietary Supplementation of Astaxanthin and Sesamin on Daily Fatigue: A Randomized, Double-Blind, Placebo-Controlled, Two-Way Crossover Study. Nutrients. 2018 Feb 28;10(3):281. doi: 10.3390/nu10030281. PMID 29495607
- [Background] Wilson LM, Tharmarajah S, Jia Y, Semba RD, Schaumberg DA, Robinson KA. The Effect of Lutein/Zeaxanthin Intake on Human Macular Pigment Optical Density: A Systematic Review and Meta-Analysis. Adv Nutr. 2021 Dec 1;12(6):2244-2254. doi: 10.1093/advances/nmab071. PMID 34157098